CLINICAL TRIAL: NCT03435575
Title: BOOSTH: Serious Gaming in Combination With Physical Activity Promotion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion rate not reached and due to the COVID-19 pandemic not enough follow up measurements of the included participants.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL61033.000.17
Record Dates: First submitted 2018-01-29; First posted 2018-02-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Physical Activity; Serious Game; Childhood Obesity; Overweight and Obesity
Keywords: physical activity; serious game; childhood obesity
MeSH Terms: conditions — Motor Activity; Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Intervention and control group parallel
Masking Description: Randomization into intervention or control group. Children in the intervention group will receive Boosth at the start of the study. Children in the control group will receive Boosth after the study is finished
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Children in the intervention group will receive Boosth: Boosth activity tracker, Boosth syncc app and Boosth game app
  Interventions: Device: Boosth
- Control group (No Intervention): Standard care

INTERVENTIONS:
Device: Boosth — Boosth activity tracker which measures steps
  Arms: Intervention group

SUMMARY:
Physical inactivity is considered to be one of the ten principal risk factors for death worldwide. Children need to perform one hour of daily moderate-to-vigorous intensity physical activity whereof at least twice a week these activities are of vigorous intensity. In 2010, the percentage of 4-11 year-old normoactive Dutch children was approximately 20%. In addition, there is a dose-response relationship between BMI by sex and physical activity levels. Previous interventions that aimed to increase childhood physical activity produced small to negligible effects. One possible explanation is that individuals were not intrinsically motivated towards PA during the intervention period. Children spend a substantial amount of their time behind a game consule. There are a number of applications that motivate increase in PA in a fun way through engaging individuals in games that mix real and computing worlds. These games became known as serious games. In this study we want to investigate if the incorporation of a serious game BOOSTH in combination with an activity tracker to stimulate physical activity behaviour in overweight/ obese children.

DETAILED DESCRIPTION:
The investigational treatment consists of regular COACH care and the BOOSTH physical activity intervention. Children in the intervention group will start with the physical activity intervention. The child will receive the BOOSTH activity tracker. The child (under supervision of their parents) needs to download the BOOSTH sync app and the BOOSTH game app. Therefore it is important that the child or their parents have a device with Bluetooth. The investigators create a login account for the child. After installing the apps, the activity tracker measures step counts which are translated into activity points. These activity points will be used to unlock levels in the BOOSTH game app. The child synchronizes their activity points, with Bluetooth connection, in the BOOSTH sync app and immediately the child could open the BOOSTH game app to play a level in the game. The child needs seven green lights (corresponding to 30 minutes of performed physical activity) to unlock a level in the game. The first four levels are for free, to gain interests of the child, but thereafter the child needs to be physically active to unlock the rest of the levels in the game. The intervention consists of a combination of supporting strategies: • BOOSTH game: it is a reward based game since the child needs to perform physical activity to unlock a level in the game. The BOOSTH game is a jump and run game. • Lights on the activity tracker: the child will be stimulated to promote physical activity by using green lights on the activity tracker. The more performed physical activity, the more green lights on the activity tracker (maximum of seven green lights). When the maximum is reached the child could use the activity points to unlock a level in the game. • Group system: a special COACH group (in the BOOSTH game app) will be created. Children can compare their scores with each other and challenge each other to gain more activity points. • Every week the child receives a reminder (by email or phone) to promote physical activity. Every week the researcher will download the BOOSTH data. Individual adjustments and encouragement could be made based on results of the data. • The medical doctor (MD) will stimulate physical activity behavior during regular COACH visits and promote the use of BOOSTH The intervention duration is 6 months. Measurements will be performed at baseline, 3-, 6- and twelve months after the start.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls, aged between 8 and 12 years (at time of inclusion)
* Overweight or obesity according to IOTF criteria Are enrolled in the COACH program
* Have access to a technological device (i.e. tablet, iPad, phone) with bluetooth option (to synchronize activity points and playing the BOOSTH game)

Exclusion Criteria:

* Children who are suffering from any musculoskeletal condition that would prevent the subject from performing PA.
* Children who already participate in another PA intervention (children who are attending COACH Sports lessons will be excluded)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
change in moderate to vigorous physical activity (min/day) | 1 week weartime at baseline, 3, 6 and 12 months
  moderate to vigorous physical activity (min/day) as measured with the Actigraph accelerometer

SECONDARY OUTCOMES:
Change in step count | up to 6 months
  Daily step count via Boosth activity tracker
Change in physical activity behaviour | up to 12 months
  Subjective physical activity behaviour via Baecke questionnaire. BAECKE (for children) will be used to assess the amount of habitual PA ranging from 1 (lowest activity) to 5 (highest activity). Physical activity at school, during leisure time and organized sports will be asked.
Anthropometry | up to 12 months
  Weight (kg) and height (cm) will be combined to report BMI in kg/m^2
Body composition | up to 12 months
  Fat Mass and Fat Free Mass via Bodpod measurement
Energy Expenditure | up to 6 months
  Energy expenditure as measured with indirect calorimetrie
Screentime | up to 12 months
  Screentime as measured with questionnaire. Subjects and their parents will report the average hours per day (weekday and weekend day) of screen-time (hours/day). Screen-time are activities like watching T.V., use of computer, playing videogames and the use of social media like Facebook or Instagram. Self-reported screen time will be reported separately for weekday and weekend day assessed with the following questions: 'How many hours a day during the last 4 weeks you watched TV on a normal weekday/weekend?' and 'How many hours a day during the last 4 weeks have you played console games or used a computer for your free time activities on a normal weekday/weekend? Possible responses are: 'not at all', '0.5 hours per day', 'one hour per day', '2 hours per day', '2.5 hours per day', '3 hours per day', '3.5 hours per day', '4 hours or more per day'. Total screen time was calculated by summing minutes spent in TV watching and computer use.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vreugdenhil, Dr, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No